CLINICAL TRIAL: NCT03526783
Title: A Comparison of the Mini/One Anastomosis-Gastric Bypass and Roux-en-Y Gastric Bypass for Conversion of Failed Sleeve Gastrectomy
Brief Title: MGB/OAGB Versus RYGB After Failed Sleeve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, MD, Senior Consultant, Principal Investigator, Sana Klinikum Offenbach
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF 3/2018
Record Dates: First submitted 2018-04-23; First posted 2018-05-16 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Obesity
Keywords: Obesity Surgery; Failed Sleeve Gastrectomy; Roux-en-Y gastric bypass; Mini/One anastomosis gastric bypass
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Failed sleeve gastrectomy - RNYGB (Other): Intervention: Roux en Y gasric bypass (RNYGB)
  Interventions: Procedure: Roux en Y gastric bypass
- Failed sleeve gastrectomy - MGB/OAGB (Other): Inervention: Mini/One anastomosis gasic bypass (MGB/OAGB)
  Interventions: Procedure: Mini/One anastomosis gastric bypass

INTERVENTIONS:
Procedure: Roux en Y gastric bypass — Laparoscopic Roux en Y gastric bypass (150 cm alimentary limb, 50 cm biliopancreaty limb)
  Other Names: RNYGB
  Arms: Failed sleeve gastrectomy - RNYGB
Procedure: Mini/One anastomosis gastric bypass — Laparoscopic Mini/One anastomosis gastric bypass (200 cm biliopancreatic limb)
  Other Names: MGB/OAGB
  Arms: Failed sleeve gastrectomy - MGB/OAGB

SUMMARY:
Sleeve Gastrectomy is the most performed bariatric procedure worldwide. But a growing number of data documents that some patients have to be surgical revised due to weight regain or gastro-esophageal reflux disease.

This study elaborates weather Roux-en-Y gastric bypass (RYGB) or Mini/One anastomosis gastric bypass (MGB/OAGB) is a better second step procedure after failed sleeve gastrectomy.

DETAILED DESCRIPTION:
All patients who underwent RYGB or MGB/OAGB between October 2014 and December 2016 after failed sleeve gastrectomy will be recorded and analyzed in relation to weight loss, intra- and postoperative complications (Clavien-Dindo) and postoperative morbidity up to one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients with failed sleeve due to

* weight regain
* weight loss failure
* gastro-esophageal reflux disease Grade B

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 1 year follow-up
  Total Body Weight Loss in %
Weight Loss | 1 year follow-up
  Excess Weight Loss in %

SECONDARY OUTCOMES:
Perioperative Complications | up to 30 days postsurgery
  Perioperative Complications (Clavin-Dindo)
Postoperative Morbidity | 1 year follow-up
  Postoperative Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Chiappetta, MD, Principal Investigator — Sana Klinikum Offenbach
Locations (1):
- Sana Klinikum Offenbach, Offenbach, Offenbach Am Main, Germany

IPD SHARING:
Plan to Share IPD: No
Anonymous data will be published.

REFERENCES:
- [Result] Almalki OM, Lee WJ, Chen JC, Ser KH, Lee YC, Chen SC. Revisional Gastric Bypass for Failed Restrictive Procedures: Comparison of Single-Anastomosis (Mini-) and Roux-en-Y Gastric Bypass. Obes Surg. 2018 Apr;28(4):970-975. doi: 10.1007/s11695-017-2991-0. PMID 29101719
- [Result] Sarela AI, Dexter SP, O'Kane M, Menon A, McMahon MJ. Long-term follow-up after laparoscopic sleeve gastrectomy: 8-9-year results. Surg Obes Relat Dis. 2012 Nov-Dec;8(6):679-84. doi: 10.1016/j.soard.2011.06.020. Epub 2011 Jul 20. PMID 21890430
- [Result] Felsenreich DM, Kefurt R, Schermann M, Beckerhinn P, Kristo I, Krebs M, Prager G, Langer FB. Reflux, Sleeve Dilation, and Barrett's Esophagus after Laparoscopic Sleeve Gastrectomy: Long-Term Follow-Up. Obes Surg. 2017 Dec;27(12):3092-3101. doi: 10.1007/s11695-017-2748-9. PMID 28593484
- [Result] Weiner RA, Theodoridou S, Weiner S. Failure of laparoscopic sleeve gastrectomy--further procedure? Obes Facts. 2011;4 Suppl 1(Suppl 1):42-6. doi: 10.1159/000327343. Epub 2011 Apr 4. PMID 22027290
- [Result] Casillas RA, Um SS, Zelada Getty JL, Sachs S, Kim BB. Revision of primary sleeve gastrectomy to Roux-en-Y gastric bypass: indications and outcomes from a high-volume center. Surg Obes Relat Dis. 2016 Dec;12(10):1817-1825. doi: 10.1016/j.soard.2016.09.038. Epub 2016 Oct 4. PMID 27887931
- [Result] Disse E, Pasquer A, Espalieu P, Poncet G, Gouillat C, Robert M. Greater weight loss with the omega loop bypass compared to the Roux-en-Y gastric bypass: a comparative study. Obes Surg. 2014 Jun;24(6):841-6. doi: 10.1007/s11695-014-1180-7. PMID 24442421